CLINICAL TRIAL: NCT06641076
Title: A Phase 3, Parallel-group, Randomized, Double-blind, 3-arm, Placebo-controlled, Multicenter Study to Investigate the Efficacy and Safety of Subcutaneous Sonelokimab in Male and Female Participants Aged 18 Years and Over With Active Psoriatic Arthritis Who Are Naive to Biologic DMARDs
Brief Title: Evaluation of Sonelokimab in Patients With Active Psoriatic Arthritis Naive to Biologic Disease-Modifying Antirheumatic Drug
Acronym: IZAR-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: MoonLake Immunotherapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M1095-PSA-301
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — sonelokimab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- sonelokimab dose with an induction regimen (Experimental): Subjects randomized to this arm will receive sonelokimab subcutaneously (SC) as an induction regimen of 4 doses, followed by sonelokimab SC every 4 weeks maintenance dosing starting at Week 8.
  Interventions: Drug: Sonelokimab
- sonelokimab dose without an induction regimen (Experimental): Subjects randomized to this arm will receive sonelokimab subcutaneously every 4 weeks.
  Interventions: Drug: Sonelokimab
- Placebo (Placebo Comparator): Subjects randomized to this arm will receive placebo subcutaneously.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sonelokimab — Randomized treatment, parallel-group
  Arms: sonelokimab dose with an induction regimen; sonelokimab dose without an induction regimen
Drug: Placebo — Randomized treatment, parallel-group
  Arms: Placebo

SUMMARY:
This is a study to demonstrate the clinical efficacy and safety of sonelokimab administered subcutaneously compared with placebo in the treatment of adult patients with active psoriatic arthritis who are naive to biologic disease-modifying antirheumatic drug therapy.

DETAILED DESCRIPTION:
M1095-PSA-301 is a Phase 3, multicenter, randomized, parallel-group, double-blind, 3-arm, placebo-controlled study to investigate the efficacy and safety of sonelokimab 60 mg every 4 weeks (with and without an induction regimen) versus placebo in adults with active psoriatic arthritis who are naive to biologic disease-modifying antirheumatic drug therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be ≥18 years of age .
2. Participants have a confirmed diagnosis of psoriatic arthritis (PsA) per the 2006 Classification for Psoriatic Arthritis (CASPAR) criteria with symptoms for ≥6 months before the Screening Visit.
3. Participants have active disease (defined by a 68 tender joint count [TJC68] of ≥3 and a 66 swollen joint count [SJC66] of ≥3).
4. Participants have current active plaque psoriasis (PsO) or a dermatologist-confirmed history of plaque PsO.
5. Participants test negative for both rheumatoid factor and anti-cyclic citrullinated peptide at the Screening Visit.

Exclusion Criteria:

1. Participants with a known hypersensitivity to sonelokimab or any of its excipients.
2. Participants who have a diagnosis of chronic inflammatory conditions other than PsO or PsA.
3. Participants with a diagnosis of inflammatory bowel disease.
4. Participants who have experienced a period of ≥3 consecutive weeks of unexplained diarrhea in the 24 weeks before the Baseline Visit.
5. Participants who have an established diagnosis of arthritis mutilans.
6. Previous exposure to sonelokimab.
7. Participants who have ever received any biologic immunomodulating agents for PsA or PsO, whether investigational or approved.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 960 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Response rate of participants achieving at least a 50% improvement in the American College of Rheumatology criteria (ACR50) | Week 16
  Proportion of participants achieving ACR50

SECONDARY OUTCOMES:
Response rate of participants achieving at least 20% improvement in the American College of Rheumatology criteria (ACR20) | Week 16
  Proportion of participants achieving ACR20
Response rate of participants achieving Minimal Disease Activity (MDA) | Week 16
  Proportion of participants achieving MDA
Health Assessment Questionnaire- Disability Index (HAQ-DI) | Week 16
  Change in HAQ-DI from baseline
Psoriasis Area and Severity Index (PASI90) | Week 16
  Proportion of participants achieving a decrease of ≥90% in the PASI90 response at Week 16 in the subgroup of participants with psoriasis (PsO) involving ≥3% body surface area at baseline
Short- form-36 (SF-36) Physical Component Summary (PCS) | Week 16
  Change from Baseline in SF-36 PCS at Week 16
van der Heijde modified Total Sharp Score (vdHmTSS) | Week 16
  Change from Baseline to Week 16 in joint/bone structural damage (vdHmTSS)

CONTACTS AND LOCATIONS:
Locations (122):
- United States (28):
  - Clinical Site, Avondale, Arizona
  - Clinical Site, Chandler, Arizona
  - Clinical Site, Flagstaff, Arizona
  - Clinical Site, Mesa, Arizona
  - Clinical Site, Phoenix, Arizona
  - Clinical Site, Scottsdale, Arizona
  - Clinical Site, Tucson, Arizona
  - Clinical Site, San Diego, California
  - Clinical Site, Upland, California
  - Clinical Site, Avon Park, Florida
  - Clinical Site, Clearwater, Florida
  - Clinical Site, Hialeah, Florida
  - Clinical Site, Tampa, Florida
  - Clinical Site, Springfield, Illinois
  - Clinical Site, Lake Charles, Louisiana
  - Clinical Site, Baltimore, Maryland
  - Clinical Site, Grand Blanc, Michigan
  - Clinical Site, Leland, North Carolina
  - Clinical Site, Salisbury, North Carolina
  - Clinical Site, Statesville, North Carolina
  - Clinical Site, Middleburg Heights, Ohio
  - Clinical Site, Portland, Oregon
  - Clinical Site, Memphis, Tennessee
  - Clinical Site, Allen, Texas
  - Clinical Site, Colleyville, Texas
  - Clinical Site, Lubbock, Texas
  - Clinical Site, Plano, Texas
  - Clinical Site, Beckley, West Virginia
- Bulgaria (5):
  - Clinical Site, Pleven
  - Clinical Site, Plovdiv
  - Clinical Site, Rousse
  - Clinical Site, Sofia
  - Clinical Site, Stara Zagora
- Canada (4):
  - Clinical Site, Calgary
  - Clinical Site, Trois-Rivières
  - Clinical Site, Waterloo
  - Clinical Site, Winnipeg
- Croatia (2):
  - Clinical Site, Rijeka
  - Clinical Site, Zagreb
- Czechia (6):
  - Clinical Site, Brno
  - Clinical Site, Břeclav
  - Clinical Site, Ostrava
  - Clinical Site, Prague
  - Clinical Site, Studénka
  - Clinical Site, Zlín
- Estonia (2):
  - Clinical Site, Tallinn
  - Clinical Site, Tartu
- Clinical Site, Kuopio, Finland
- France (8):
  - Clinical Site, Cahors
  - Clinical Site, Caluire-et-Cuire
  - Clinical Site, Échirolles
  - Clinical Site, Montpellier
  - Clinical Site, Narbonne
  - Clinical Site, Nice
  - Clinical Site, Rouen
  - Clinical Site, Tours
- Georgia (2):
  - Clinical Site, Kutaisi
  - Clinical Site, Tbilisi
- Germany (7):
  - Clinical Site, Bad Bentheim
  - Clinical Site, Berlin
  - Clinical Site, Erlangen
  - Clinical Site, Hamburg
  - Clinical Site, Herne
  - Clinical Site, Munich
  - Clinical Site, München
- Greece (2):
  - Clinical Site, Athens, Attica
  - Clinical Site, Heraklion
- Hungary (10):
  - Clinical SIte, Budapest
  - Clinical Site, Budapest
  - Clinical Site, Debrecen
  - Clinical Site, Gyula
  - Clinical Site, Hódmezővásárhely
  - Clinical Site, Kalocsa
  - Clinical Site, Kistarcsa
  - Clinical Site, Nyíregyháza
  - Clinical Site, Székesfehérvár
  - Clinical Site, Veszprém
- Latvia (2):
  - Clinical Site, Ādaži
  - Clinical Site, Riga
- Lithuania (2):
  - Clinical Site, Kaunas
  - Clinical Site, Šiauliai
- Poland (21):
  - Clinical Site, Bialystok
  - Clinical Site, Bydgoszcz
  - Clinical Site, Bytom
  - Clinical Site, Częstochowa
  - Clinical Site, Dąbrówka
  - Clinical Site, Elblag
  - Clinical Site, Gdynia
  - Clinical Site, Krakow
  - Clinical Site, Lodz
  - Clinical Site, Lublin
  - Clinical Site, Nadarzyn
  - Clinical Site, Nowa Sól
  - Clinical Site, Olsztyn
  - Clinical Site, Poznan
  - Clinical Site, Siedlce
  - Clinical Site, Sochaczew
  - Clinical Site, Swidnica
  - Clinical Site, Torun
  - Clinical Site, Warsaw
  - Clinical Site, Wołomin
  - Clinical Site, Wroclaw
- Portugal (3):
  - Clinical SIte, Braga
  - Clinical Site, Braga
  - Clinical Site, Lisbon
- Romania (2):
  - Clinical Site, Bucharest
  - Clinical Site, Timișoara
- Serbia (2):
  - Clinical Site, Belgrade
  - Clinical Site, Novi Sad
- Slovakia (4):
  - Clinical Site, Košice
  - Clinical Site, Martin
  - Clinical Site, Poprad
  - Clinical Site, Rimavská Sobota
- Spain (9):
  - Clinical Site, A Coruña
  - Clinical Site, Bilbao
  - Clinical Site, Castelló
  - Clinical Site, Madrid
  - Clinical Site, Málaga
  - Clinical Site, Sabadell
  - Clinical Site, Santiago de Compostela
  - Clinical Site, Seville
  - Clinical Site, Valencia